CLINICAL TRIAL: NCT06196775
Title: A Single-arm, Single-center, Phase II Clinical Trial of Cadonilimab (Anti PD-1/CTLA-4) Combined With AK112 (Anti VEGF/PD-1) as Second-line Therapy in Patients With Unresectable Locally Advanced, Recurrent or Metastatic Hepatocellular Carcinoma
Brief Title: A Study of Cadonilimab Combined With AK112 as Second-line Therapy in Patients With Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, Director, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-042
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: cadonilimab (anti PD-1/CTLA-4 bispecific antibody); AK112 ( anti VEGF/PD-1 bispecific antibody)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104+AK112 (Experimental)
  Interventions: Biological: AK104+AK112

INTERVENTIONS:
Biological: AK104+AK112 — Cadonilimab (AK104): 10mg/kg or 15mg/kg Q6W iv D8 (dose choosing depends on the outcome of the dose climb stage) AK112: 20mg/kg Q3W iv D1 Eligible patients will receive AK104 plus AK112 until disease progression or withdrawn ICF or death, whichever comes first.

SUMMARY:
To evaluate the efficacy and safety of cadonilimab combined with AK112 as second-line therapy in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed HCC
* Age 18-75 years old
* ECOG PS 0-1
* Child Pugh A-B7
* Patients who progressed on first-line standard system therapy (immunotherapy combined with Anti-angiogenesis targeting regimen) or with intolerable toxicity
* At least one measurable lesion (RECIST 1.1)
* Enough organ and bone marrow function
* Expected survival time≥12 weeks
* Sign a written informed consent and be able to comply with the visit and related procedures required by the study protocol

Exclusion Criteria:

* Severe complications due to primary liver disease
* No prior systemic therapy for advanced or metastatic primary hepatocellular carcinoma
* Malignant diseases other than primary hepatocellular carcinoma were diagnosed within 5 years prior to first administration
* Previous treatment with drugs that synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137)
* Autoimmune immune disease
* History of HIV
* Prognent women
* The presence of any serious or uncontrolled systemic disease
* Medical history or evidence of disease that may interfere with the test results, prevent participants from participating fully in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers that there are other potential risks that are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | From the first drug administration up to two years
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate | From the first drug administration up to two years
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.
Disease control Rate | From the first drug administration up to two years
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Overall survival | From the first drug administration up to two years
  Defined as the time between the first dose to death due to any causes.
Incidence of Adverse Events | From the first drug administration to within 90 days for the last dose
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Hospital, Harbin, China